CLINICAL TRIAL: NCT02837796
Title: Effects of Trans-Obturator Tape outside-in Versus Inside-out Procedure for Stres Urinary Incontinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Bakirkoy Maternity and Children Diseases Hospital (Other Government)
Responsible Party: Principal Investigator, Osman Aşıcıoğlu, medical doctor, Istanbul Bakirkoy Maternity and Children Diseases Hospital
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: Asıcıoglu09
Record Dates: First submitted 2016-07-12; First posted 2016-07-20 (Estimated); Last update posted 2016-07-20 (Estimated); Status verified 2016-07

CONDITIONS: Quality of Life; Sexual Dysfunction
MeSH Terms: conditions — Sexual Dysfunction, Physiological | interventions — Suburethral Slings

ARMS (2):
- inside-outside group (Active Comparator): inside-out transobturator tape approach
  Interventions: Procedure: transobturator tape
- outside-inside group (Active Comparator): outside-in transobturator tape approach
  Interventions: Procedure: transobturator tape

INTERVENTIONS:
Procedure: transobturator tape

SUMMARY:
The investigators think that the two techniques of TOT (inside-out and outside-in) procedures both statistically improve the sexual functions, psychosocial state and quality of life after the surgery. Additionally postoperative physical and behavioral-emotional scores in PISQ-12 were statistically more increase in inside-out group than the outside-in group.

ELIGIBILITY:
Inclusion Criteria:

* pure urodynamic SUI
* sexual active before and 2 months after the surgery
* married or single
* aged over 20
* have cured after TOT operation

Exclusion Criteria:

* preoperative or postoperative detrusor disfunction
* previous history of malignancy
* prior vaginal surgery
* a partner with sexual incapabilities
* a concomitant gynecologic disorder
* patients with pelvic organ prolapse over stage II
* pelvic radiotherapy and a history of psychological diseases
* participants who had no sexual activity with in the past two months

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2013-09; Primary Completion 2014-09 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
postoperative differences at emotional-behavioral PISQ-12 score | 1 year
postoperative differences at physical PISQ-12 score | 1 year

REFERENCES:
- [Result] Asoglu MR, Selcuk S, Cam C, Cogendez E, Karateke A. Effects of urinary incontinence subtypes on women's quality of life (including sexual life) and psychosocial state. Eur J Obstet Gynecol Reprod Biol. 2014 May;176:187-90. doi: 10.1016/j.ejogrb.2014.02.008. Epub 2014 Feb 15. PMID 24630299